CLINICAL TRIAL: NCT06333873
Title: Validation of Standardized Tasks and Questionnaires to Evaluate and Understand the Impact of Age-related Macular Degeneration on Daily Living Activitie
Brief Title: Impact of Age-related Macular Degeneration on Daily Living Activitie
Acronym: AMDAY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier National d'Ophtalmologie des Quinze-Vingts (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: P22-09
Record Dates: First submitted 2024-01-26; First posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Patient Reported Outcome Measures

STUDY DESIGN:
Intervention Model Description: Prospective, longitudinal, interventional, exploratory, non-randomised, single-centre study including healthy volunteers and patients with AMD
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Patients with early-stage AMD (Other): 30Patients with early-stage AMD
  Interventions: Other: patient-reported outcome
- Patients with intermediate-stage AMD (Other): 30 with intermediate-stage AMD
  Interventions: Other: patient-reported outcome
- 30 healthy volunteers (Other): Without AMD risk
  Interventions: Other: patient-reported outcome
- 30 healthy volunteers with central microdrusens (at risk of developing AMD) (Other): with central microdrusens (at risk of developing AMD)
  Interventions: Other: patient-reported outcome

INTERVENTIONS:
Other: patient-reported outcome — Performance of real-life tests and tasks

SUMMARY:
The complex and variable course of age-related diseases makes it all the more necessary to carry out personalised, reasoning-based examinations to improve the personalised assessment and management of AMD. However, functional assessment of AMD is most often based solely on visual acuity, and classifications of AMD are based solely on structural markers. There is therefore a need to improve the detection and functional assessment of this vision-threatening eye disease, by complementing and extending the standard assessments of clinical outcomes (COA)

DETAILED DESCRIPTION:
Prospective, longitudinal, interventional, exploratory, non-randomised, single-centre study, including healthy volunteers and patients with Age-Related Macular Degeneration

ELIGIBILITY:
Inclusion Criteria:

* General criteria for healthy volunteers and AMD patients:

  * Male / Female participant,
  * Age ≥ 50 at inclusion,
  * Able and willing to provide written informed consent and comply with the study protocol, visits and assessments,
  * Quality of AO imaging as assessed by rtx1 camera, ● deemed adequate according to the study physician,
  * Membership of a social security scheme or beneficiary of such a scheme.
* Specific criteria for the AMD group:

  * Geriatric Depression Scale (GDS) questionnaire score ≤ 10 A COGEVIS questionnaire score ≥ 24/30
  * Visual acuity greater than 4/10ths
* General criteria for healthy volunteers:

  * No detectable visual pathologies
  * Best monocular visual acuity (corrected to 100% of the contrast) ≥ 8/10ths before age 70 and ≥ 6/10ths after.
  * MMSE score ≥ 20
* Specific criteria for the group of healthy volunteers with central microdrusens:

  * No detectable visual pathologies other than the presence of central microdrusens.
  * Best monocular visual acuity (corrected to 100% contrast) ≥ 8/10th before age 70 and ≥ 6/10th after.
  * MMSE score ≥ 20

Exclusion Criteria:

* Pregnant, parturient or breast-feeding women,
* Subjects taking medication likely to cause motor, visual, vestibular or cognitive disorders (PSA, neuroleptics, etc.) or who could interfere with the study examinations cannot be included in this study,
* Environmental opacity or eye movement disorders (nystagmus) which, in the opinion of the investigator, interfere with the quality of retinal imaging data.
* Any concomitant intraocular condition in the study eye (e.g. glaucoma or cataract) that, in the opinion of the investigator, would require surgical intervention during the study to prevent or treat vision loss that may result from this condition or affect the interpretation of study results,
* Known systemic disease which, in the opinion of the investigator, would preclude active participation in the study,
* Participation in any other therapeutic study evaluating a drug,
* Cognitively impaired subjects, illiterate subjects and subjects who do not speak the national language.
* Subjects with dyslexic reading disorders,
* Subjects subject to a reinforced protection measure or legal safeguard (curatorship, guardianship).

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2029-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Validity of criteria | 26 month
  Number of patients with capacity of discrimintaion compared to healthy volunteers.
  ROC (receiver operating characteristic curve), which illustrates the diagnostic capacity of a binary classification system as a function of the variation in its discrimination threshold. The ROC curve is created by plotting the rate of true positives versus the false-positive rate for different thresholds. The index used to characterize a test's of a test is the air under the curve
Validity of content | 26 month
  number of paticipants with capacity to execute questionnaires and daily real-life task
Reproducibility of results | 26 month
  Number of patients able to reproduce the same performance tests

CONTACTS AND LOCATIONS:
Overall Officials: Michel PAQUES, Pr, Principal Investigator — centre Hospitalier Nationald'Ophtalmologie